CLINICAL TRIAL: NCT05188339
Title: Compare Effectiveness and Safety Utilizing 4% Sodium Citrate vs. Heparin as a Lock Solution in Central Venous Hemodialysis Catheter Among Hemodialysis Patients
Brief Title: The Effectiveness and Safety of 4% Sodium Citrate as a Lock Solution in Central Venous Hemodialysis Catheter
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB No.: 202100060A3
Record Dates: First submitted 2021-12-06; First posted 2022-01-12 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-04

CONDITIONS: Central Venous Catheter Thrombosis; Renal Dialysis
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis | interventions — Sodium Citrate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 4% sodium citrate group (Experimental): Dose of 4% sodium citrate is also according to catheter lumen (LVR) instilled into each lumen of catheter after HD session, eg. 1.6 cc/lumen for LV R 1.6, 1.8 cc/lumen for LVR 1.8.
  Interventions: Drug: 4% sodium citrate
- heparin group (Active Comparator): Heparin dosage is based on volume ratio in catheter lumen (LVR) after each HD session, eg. 8000u/lumen in 1.6 LVR, 9000u/lumen in LVR 1.8.
  Interventions: Drug: heparin group

INTERVENTIONS:
Drug: 4% sodium citrate — Dose of 4% sodium citrate is also according to catheter lumen (LVR) instilled into each lumen of catheter after HD session, eg. 1.6 cc/lumen for LV R 1.6, 1.8 cc/lumen for LVR 1.8.
  A prospective, open label, control study. The content of study protocol will be posted in the HD room in the Kaohsiung Chang Gung memorial Hospital, Taiwan. After inform consent obtained, we will categorize enrolled participants randomly into two groups, 4% sodium citrate group(experimental group), heparin group(control group), respectively. The study duration is three months.
  Other Names: there is no other intervention names
  Arms: 4% sodium citrate group
Drug: heparin group — Heparin dosage is based on volume ratio in catheter lumen (LVR) after each HD session, eg. 8000u/lumen in 1.6 LVR, 9000u/lumen in LVR 1.8.
  Other Names: there is no other intervention names
  Arms: heparin group

SUMMARY:
Studies that used a dilute citrate formulation (4%) demonstrated efficacy as an anticoagulant with minimal to no risk of bleeding in HD sessions. This study will compare effectiveness and safety utilizing 4% sodium citrate vs. heparin as a lock solution in central venous hemodialysis catheter among hemodialysis patients.

DETAILED DESCRIPTION:
Vascular access is necessary for hemodialysis(HD) procedure. In normal situation, vascular access for HD is created in peripheral vessels. However, vascular catheter may be considered in patients without available peripheral vessels for vascular access. The characteristic of these patients include elderly, diabetes, not tolerant to vascular surgery etc.. Commonly, the HD catheter is inserted in the central vein in these population. Considering clotting condition, anticoagulant is indicated for catheter locking after HD session. In the past years, heparin is the most common solution to be used as locking solution. Nevertheless, heparin has a few disadvantages, such as systemic anticoagulation, thrombocytopenia, and bleeding risk. An alternative for anticoagulation in HD session is 4% sodium citrate. The effectiveness and safety of sodium citrate in HD sessions have been reported in clinical studies.

Characteristics of sodium citrate and safety profile Trisodium citrate acts locally as an anticoagulant by chelating ionized calcium in blood, resulting in the blockage of calcium-dependent clotting pathways. Studies that used a dilute citrate formulation (4%) demonstrated efficacy as an anticoagulant with minimal to no risk of bleeding in HD sessions. The advantageous effects of sodium citrate in HD catheter locking solution includes reducing frequency of catheter exchanges, reducing using of thrombolytic drugs, reducing hospitalization rates, and bacteremia. Regarding adverse effect of sodium citrate, hypocalcemia and other untoward outcomes are rare reported in the previous clinical studies

ELIGIBILITY:
Inclusion Criteria:

1. Age >=20 years
2. End-stage renal disease patients who received regular HD weekly via central venous catheter for at least 3 months in outpatient clinic in Kaohsiung Chang Gung Memorial Hospital, Taiwan

Exclusion Criteria:

1. bleeding tendency
2. on radiotherapy or chemotherapy for malignancy
3. pregnancy
4. drug allergy history to citrate
5. undefined reasons for refuted participation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
central venous catheter exchanges | 3 months
  We will record the episode of central venous catheter malfunction and central venous catheter exchanges within the period of trial and compare the incidence between two arms.

SECONDARY OUTCOMES:
events of thrombolytic drug use, bacteremia and all-cause hospitalization days. | 3 months
  We will record the episode of central venous catheter malfunction and events of thrombolytic drug use within the period of trial and compare the incidence between two arms.
  We will also compare the incidence of bacteremia and all-cause hospitalization days within these 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan